CLINICAL TRIAL: NCT03974581
Title: Pharmacoinvasive Strategy vs. Percutaneous Coronary Intervention in ST-Elevation Myocardial Infarction: A Prospective, Real-World Registry in a Large Geographical Area
Brief Title: Pharmacoinvasive Strategy vs. Primary PCI in STEMI: A Prospective Registry in a Large Geographical Area
Acronym: PHASE-MX
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Diego Araiza-Garaygordobil, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: PT-19-021
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Myocardial Infarction, Acute
Keywords: pharmacoinvasive strategy; Mexico; registry
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacoinvasive strategy: Patients whom received pharmacoinvasive strategy (fibrinolysis and subsequently PCI) as reperfusion treatment.
  Interventions: Other: Primary percutaneous coronary intervention
- Primary PCI: Patients whom primary PCI as reperfusion treatment.
  Interventions: Other: Pharmacoinvasive strategy

INTERVENTIONS:
Other: Primary percutaneous coronary intervention — Patient receives primary percutaneous coronary intervention as part of his treatment; decision to allocate by treating physician.
  Other Names: Primary PCI
  Groups: Pharmacoinvasive strategy
Other: Pharmacoinvasive strategy — Patient receives primary fibrinolysis and subsequent coronary angiography (pharmacoinvasive strategy) as part of his treatment; cases with failed fibrinolysis are scheduled for immediate rescue PCI. Decision to allocate by treating physician.
  Groups: Primary PCI

SUMMARY:
For patients presenting with ST-elevation myocardial infarction (STEMI), immediate and timely reperfusion treatment is essential. Pharmacoinvasive strategy (PIs) exploits the widespread availability of fibrinolysis and its early administration to restore some degree of myocardial blood flow, coupled with the complete restoration of the culprit coronary artery patency that can be obtained with subsequent angioplasty. Several trials have demonstrated the efficacy and safety of PIs when compared with PPCI; however, real-world data is lacking, especially in developing countries.

The aim of this study was to compare safety and efficacy of PIs with PPCI in real-world patients with STEMI presenting to large geographical area.

DETAILED DESCRIPTION:
For patients presenting with ST-elevation myocardial infarction (STEMI), immediate and timely reperfusion treatment is essential. The optimal choice between primary percutaneous coronary intervention (PPCI) and intravenous thrombolytic agents depends upon the timeliness of effective delivery, as well as the total ischemic time. While PPCI is widespread available in the USA and Europe, limited resources and lack of infrastructure means that patients with STEMI in low- and middle-income countries (LMICs) receive significantly less reperfusion therapy, and when they do, they are more prone to receive thrombolytic agents.

Pharmacoinvasive strategy (PIs) exploits the widespread availability of fibrinolysis and its early administration to restore some degree of myocardial blood flow, coupled with the complete restoration of the culprit coronary artery patency that can be obtained with subsequent angioplasty. Several trials have demonstrated the efficacy and safety of PIs when compared with PPCI; however, real-world data is lacking. The aim of this study was to compare safety and efficacy of PIs with PPCI in real-world patients with STEMI presenting to large geographical area.

PHASE-Mx study is a prospective, real-world registry including patients with STEMI finally treated at a large cardiovascular center. In brief, patients aged 18-99 years old with the diagnosis of STEMI whom received either PI or PPCI during the first 12 hours since symptom onset were included. Patients could have a first medical contact directly at the study center or in one of other 60 hospitals along the STEMI network. Patients with a discharge diagnosis other than STEMI were excluded. Four of the investigators recorded the study data at admission and during hospital stay. Main efficacy outcome will be the composite of cardiovascular death, cardiogenic shock, reinfarction or stroke. Main safety outcome will include rates of major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-99 years old, with the diagnosis of STEMI whom received either PI or PPCI during the first 12 hours since symptom onset. Patients could have a first medical contact directly at the study center or in one of other 60 hospitals along the STEMI network.

Exclusion Criteria:

* Patients with a discharge diagnosis other than STEMI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI presenting to a primary reperfusion center in the metropolitan area of Mexico City.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Composite of cardiovascular mortality + cardiogenic shock + reinfarction + stroke. | 30-days follow-up.
  Main efficacy combined outcome including cardiovascular mortality, cardiogenic shock, reinfarction and stroke.

SECONDARY OUTCOMES:
Major bleeding | Major bleeding during a 30-days follow-up.
  Major bleeding during a 30-days follow-up.
All-cause mortality | 1-year follow up.
  All cause mortality at 1-year follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiología "Ignacio Chavez", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided